CLINICAL TRIAL: NCT02095119
Title: Phase I-II Study of Palliative Treatment With Nimotuzumab as a Second, Third Line or More of Treatment for Advanced or Metastatic Cervical Cancer
Brief Title: A Monoclonal Antibody, Nimotuzumab, as Treatment for Recurrent or Metastatic Cervical Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Cancerología (Other Government)
Responsible Party: Principal Investigator, Dr. Lucely Cetina Pérez, MsC, MD, National Institute of Cancerología
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INCAN/CC/130/09
Record Dates: First submitted 2014-02-17; First posted 2014-03-24 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-04

CONDITIONS: Uterine Cervical Cancer
Keywords: Uterine cervical cancer; Palliative; Treatment; Monoclonal antibody; Nimotuzumab
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — nimotuzumab; Cisplatin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Nimotuzumab — Monoclonal antibody Nimotuzumab will be administered alone at a 200mg dose weekly during the first 4 weeks. Posteriorly it will be administered with a maintenance dose of 200 mg every 2 weeks in combination with chemotherapeutic agents Cisplatin in patients with good renal function or Gemcitabine in patients with kidney failure data until exclusion or death occurs. The administration will be intravenously in 250 ml of saline solution in a time period of 30 minutes.
Drug: Cisplatin — Cisplatin will be administered at a calculated dose of 50mg/m2/BSA every 21 days as concomitant therapy to Nimotuzumab, until 6 cycles are completed, exclusion or death occurs, only in patients whose creatinine clearance as defined by the Cockcroft-Gault equation is >/= 60. The administration form will be intravenously.
Drug: Gemcitabine — Gemcitabine will be administered at a calculated dose of 800 mg/m2/BSA every 21 days as concomitant therapy to Nimotuzumab, until 6 cycles are completed, exclusion or death occurs, in patients with kidney failure data(Creatinine clearance as defined by the Cockcroft -Gault equation < 60). The administration form will be intravenously.
Procedure: CT Scan — A CT Scan will be performed in all patients prior to the beginning of treatment to assess any measurable tumor found by this method. The CT Scan will be repeated once the patient completes the induction phase with Nimotuzumab (4 once a week doses), when the patient has completed 3 full cycles of combination therapy with Nimotuzumab (every 2 weeks)and Gemcitabine or Cisplatin (every 21 days)and once more when the patient has completed 6 full cycles of the aforementioned therapy.

SUMMARY:
The following is an open label, non comparative, pilot study of palliative treatment as a second, third line or more of treatment in patients with recurrent, persistent or Metastatic Cervical Cancer; it has a limited sample of 15 patients with the primary goal of evaluating the response (defined as: Complete, partial or stable disease) to treatment with a Monoclonal Antibody, Nimotuzumab, on a weekly basis + CDDP 50mg/m2/BSA as a single agent every 3 weeks for patients with good renal function (Creatinine clearance => 60) or Gemcitabine 800 mg/m2/BSA in patients with renal failure (Creatinine clearance <60).

Secondary objectives consist of evaluating disease-free survival, overall survival and assess patient tolerance to treatment with Nimotuzumab.

ELIGIBILITY:
Diagnostic criteria:

* Female patients in whom a diagnosis of cervical cancer of epithelial origin has been confirmed by histologic and/or radiologic assessment.
* Said patients must be in relapse or persistency after receiving first line chemo-radiotherapy and one or more lines of palliative chemotherapy.
* Karnofsky score of 80 or more.
* A CT scan will be performed in all patients to assess measurable target lesions.
* The clinical diagnosis must be evaluated by more than clinical investigator

Inclusion Criteria:

* Patients who give their written consent of participation in this study.
* Patients with recurrent or persistent cervical-uterine cancer, with local and/or systemic disease with measurable lesions, whether by physical examination, CT Scan or MRI detected at least in the previous 6 weeks. If there is only one lesion and it is less than 10 mm in length, a biopsy confirmation is required.
* Patients currently receiving a second, third line or more of palliative chemotherapy diagnosed at least 30 days after the last chemotherapy.
* Patients with one of the following Histopathological reports: Squamous Cell Carcinoma (epidermoid carcinoma), adenocarcinoma, adenosquamous carcinoma or glassy cell carcinoma.
* Patients must be older than 18 years old.
* ECOG score no worst than 3.
* Patients with life expectancy greater than 4 weeks.
* Patients with left ventricle ejection fraction (LVEF) ≥ 50 measured by radioisotopic ventriculography.
* Patients who meet all previous criteria with previously radiated metastatic disease in the central nervous system will be included.
* Patients with normal functioning of the bone marrow and other organs as defined by the following parameters:
* Hemoglobin ≥ 9 g/L
* Leucocytes ≥ 4000/microL
* Absolute neutrophil count ≥ 1500/microL
* Platelet count ≥ 100000/microL
* Total serum Bilirubin: up to 1.5 times the normal value
* Total Proteins: Within normal limits
* AST and ALT =/< 2.5 times the normal superior limit of the institutional laboratory
* Serum creatinine: within normal limits or up to 2 mg and GFR ≥ 60ml/min calculated with the Cockcroft-Gault equation.

Exclusion Criteria:

* Pregnant or nursing mothers.
* Patients with cervical-uterine cancer with a histopathological report of: small cell carcinoma and/or neuroendocrine tumor.
* Patients currently receiving another investigational onco-specific drug.
* Patients with a history of allergy to chemical substances with similar chemical composition to that of the monoclonal antibody or chemotherapeutic agents used in this study.
* Patients with non-controlled co-morbid states such as active infections, symptomatic congestive heart failure, unstable angina, cardiac arrhythmias, uncompensated diabetes and/or psychiatric illness.
* Presence of a second tumor. With the exception of those patients who have received adequate treatment for skin carcinomas (basal or squamous).
* Previous or concomitant malignancy except non-melanoma skin carcinoma.
* Social, familiar or geographic conditions that suggest poor attachment to the study.

Discontinuation of treatment criteria:

* At the patient´s request.
* Progression of disease causing worsening of the patient´s overall status in non manageable clinical conditions, (ECOG worst than 3).
* Death.
* Discontinuation of monitoring and/or loss of patient follow-up for more than 2 months.
* Severe adverse reaction grade 4 according to CTCAE.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2008-07; Primary Completion 2013-12 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Antitumoral Response | After 4 weeks of induction therapy, and then every 3 months for a period of 2 years
  Treatment response will be evaluated according to the new International Criteria from Response Evaluation Committee in Solid Tumors (RESIST). Antitumoral response will be evaluated from patient´s inclusion after 4 weeks of induction therapy and then every 3 months until second year of follow up for each patient.

SECONDARY OUTCOMES:
Progression Free Survival | After patient´s inclusion every 3 months for a period 2 years
  Progression Free Survival will be defined as the time elapsed since the beginning of interventions until progressive disease is documented by growth of measurable lesions or new lesions on CT Scan or MRI according to the response evaluation criteria in solid tumors (JNCI 92 (3): 205-216, 2000).
Overall Survival | from patient´s inclusion until 24 months
  Patient´s survival since inclusion until death
Drug Toxicity | from patient´s inclusion every 2 weeks for a period of 2 years
  Drug toxicity will be assessed with hematologic, renal and hepatic laboratory measures as well as patient symptomatology and physical findings. Any abnormality in these parameters will be reported as an adverse event according to the Common Terminology Criteria for Adverse Events version 3.0(CTCAEV3.0, 2006)

CONTACTS AND LOCATIONS:
Overall Officials: Lucely Cetina, MD, Principal Investigator — Researcher Level D; Sergio A. Zapata, MD, Study Chair — Instituto Nacional de Cancerologia de Mexico; Roberto Jimenez, MD, Study Chair — Instituto Nacional de Cancerologia de Mexico; Tania Crombert, MD, Study Chair — Centro Molecular de La Habana; Mayra Ramos, MD, Study Chair — Centro Molecular de La Habana; Ezequiel Fuentes, MD, Study Chair — Pisa® Farmacéutica
Locations (1):
- Instituto Nacional de Cancerología, Mexico City, Federal District, Mexico

REFERENCES:
- [Derived] Cetina L, Crombet T, Jimenez-Lima R, Zapata S, Ramos M, Avila S, Coronel J, Charco E, Bojalil R, Astudillo H, Bazan B, Duenas-Gonzalez A. A pilot study of nimotuzumab plus single agent chemotherapy as second- or third-line treatment or more in patients with recurrent, persistent or metastatic cervical cancer. Cancer Biol Ther. 2015;16(5):684-9. doi: 10.1080/15384047.2015.1026483. PMID 25802932